CLINICAL TRIAL: NCT06665776
Title: A Prospective Observational Human Subject Research to Explore the HLA-A*02:01 Allele Frequency and the NY-ESO-1 Expression Status in Cancer Patients in Taiwan
Brief Title: HLA-A*02:01 Allele Frequency and the NY-ESO-1 Expression Status in Cancer Patients in Taiwan
Status: Recruiting | Type: Observational
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Other Study IDs: TCRT-HR2022
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor Malignancy
Keywords: NY-ESO-1; HLA-A*02:01; Solid tumor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective observational research to explore the frequency of Human leukocyte antigen A allele 02:01 (HLA*02:01) and the expression status of New York esophageal squamous cell carcinoma-1 (NY-ESO-1) in cancer patients in Taiwanese population.

DETAILED DESCRIPTION:
T cell receptor (TCR)-engineered T cells with high affinity to NY-ESO-1 epitope presented by HLA-A*02:01 are potential therapeutic strategy against solid tumor, which show exciting results in several clinical studies. However, the prevalence of patients expressing HLA-A*02:01 and NY-ESO-1 in Taiwanese population is still unknown. This research aims to explore the prevalence of cancer patients expressing HLA-A*02:01 and NY-ESO-1 in Taiwanese population. Eligible patients with triple-negative breast cancer, hepatocellular carcinoma, head and neck squamous cell carcinoma excluding nasopharyngeal carcinoma, Lung squamous cell cancer, synovial sarcoma, esophageal squamous cell carcinoma, cervical cancer, or ovarian cancer will be enrolled. High resolution genotyping for HLA-A*02:01 and NY-ESO-1 expression status using IHC will be assessed in all enrolled patients. The frequency of HLA-A*02:01 allele and the prevalence of NY-ESO-1 positive expression will be analysed by pooled patient population and by specific tumor type.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign an informed consent form (ICF).
2. Adult aged ≥ 18 years at the time of informed consent (or other age required by local regulations).
3. Confirmed diagnosis of any of the following solid tumor:

   1. Head and neck squamous cell carcinoma, excluding nasopharyngeal carcinoma;
   2. Hepatocellular carcinoma;
   3. Lung squamous cell carcinoma;
   4. Synovial sarcoma;
   5. Triple-negative breast cancer;
   6. Esophageal squamous cell carcinoma;
   7. Cervical cancer;
   8. Ovarian cancer
4. Patient who received standard curative or palliative therapy including but not limited to any targeted therapy based on mutation status for their cancer, or patient with advanced solid tumors for which there is no accepted therapy, standard therapies are no longer effective, or the patient refuses additional standard therapy.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
6. Body weight ≥ 50 Kg.
7. Life expectancy of ≥ 6 months.
8. Patient who agrees to provide the tumor sample for NY-ESO-1 IHC staining, from either fresh or archival tissue

Exclusion Criteria:

1. Known primary immunodeficiency (such as Severe Combined Immunodeficiency Disease or AIDS).
2. Uncontrolled intercurrent illness which is not suitable for enrollment at the discretion of the investigator, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements.
3. Currently confirmed diagnosis of at least 2 active cancers; patient who was cured of the other cancer [disease free period > 6 months] and currently has only one research targeted tumor can be enrolled.
4. Untreated or symptomatic brain metastasis.
5. History of organ transplantation or allogeneic stem cell transplantation.
6. Other conditions (e.g. previous use of any cell therapy) which are not suitable for enrollment at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed diagnosis of any of the following solid tumor:
  1. Head and neck squamous cell carcinoma, excluding nasopharyngeal carcinoma;
  2. Hepatocellular carcinoma;
  3. Lung squamous cell carcinoma;
  4. Synovial sarcoma;
  5. Triple-negative breast cancer;
  6. Esophageal squamous cell carcinoma;
  7. Cervical cancer;
  8. Ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The frequency of HLA-A*02:01 allele in patients with confirmed diagnosed solid tumor. | 1 day
  To explore the frequency of HLA-A*02:01 allele using genotyping with high resolution in all eligible patients with confirmed diagnosed solid tumor.
The prevalence of NY-ESO-1 positive expression in all tumor patients with HLA-A*02:01 allele. | 1 day
  To explore the prevalence of NY-ESO-1 positive expression using immunohistochemistry (IHC) in all patients with HLA-A*02:01 allele.

CONTACTS AND LOCATIONS:
Locations (6):
- Taiwan (6):
  - Chang Gung Memorial Hospital, Chiayi Branch, Chiayi City, Taiwan
  - Taichung Veterans General Hospital, Taichung, Taiwan
  - National Cheng Kung University Hospital, Tainan, Taiwan
  - Taipei Veterans General Hospital, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided